CLINICAL TRIAL: NCT05726305
Title: Transplantation of Uterus for Uterine infertiLIty From Living Donor or Deceased Donor
Acronym: TULIPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC20_9902_TULIPE
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Uterine Factor Infertility

STUDY DESIGN:
Intervention Model Description: Living donor versus deceased donor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live donor uterus transplantation (Experimental): Transplantation of uterus from a living donor. Immunosuppression with tacrolimus.
  Interventions: Procedure: Live donor uterus transplantation
- Deceased donor uterus transplantation (Experimental): Transplantation of uterus from a deceased brain-dead donor. Immunosuppression with tacrolimus.
  Interventions: Procedure: Deceased donor uterus transplantation

INTERVENTIONS:
Procedure: Live donor uterus transplantation — Transplantation of uterus from a living donor.
  Arms: Live donor uterus transplantation
Procedure: Deceased donor uterus transplantation — Transplantation of uterus from a deceased brain-dead donor.
  Arms: Deceased donor uterus transplantation

SUMMARY:
Patients with absolute Uterine Factor Infertility (AUFI) are infertile due to the absence of a uterus. The absence of a uterus can be either iatrogenic (hysterectomy for gynecological pathology such as cancer or for obstetric pathology such as postpartum hemorrhage with hysterectomy for hemostasis), or congenital with utero-vaginal agenesis including Mayer Rokitansky Küster Hauser syndrome (MRKH) is the most common syndrome of uterine agenesis.

Alongside the AUFI, there is Non-Absolute Uterine Factor Infertility (NAUFI) which corresponds to patients with a uterus in place but which is altered by different pathologies, most often acquired, making it unsuitable for embryonic implantation and preventing the patient to get pregnant.

Uterus Transplantation (UT) represents an interesting alternative to the treatment of AUFI and potentially NAUFI (in the event of a uterus present but unsuitable for implantation) to access parenthood, especially since it is the only proposal that allows the patient to be both the surrogate mother, the biological mother (in case of simple donation) and the legal mother.

Many animal experiments have been accelerated since the beginning of the 21st century demonstrating that uterus transplantation was technically feasible and that pregnancy was possible.

In humans, several teams have recently performed several uterus transplants and have shown that this procedure is possible whether the donor is alive or dead (state of brain death).

In France, two teams (Foch and Limoges) have developed a uterus transplantation program. One in the context of living donors and the other of a deceased donors.

At the University Hospital of Rennes, we want to offer a UT program allowing access to a living or deceased donor for women with AUFI (type 1 or 2 MRKH syndrome and hysterectomy).

DETAILED DESCRIPTION:
Methods: Sixteen UT will be performed in total in 2 parallel arms: 8 UT from a live donor and 8 UT from a deceased brain-dead donor. Patients who have no suitable live donor will be wait-listed for a deceased donor.

Phases of the UT procedure: selection, in vitro fertilization and cryopreservation of embryos, uterus retrieval from a live donor or from a deceased donor, orthotopic uterus transplantation , follow up period (12 months), embryo transfer, pregnancy, child birth via Cesarian section (2 children maximum), later graft hysterectomy.

ELIGIBILITY:
Inclusion Criteria for UT recipient:

* Patient aged 18 to 40 at the time of the UT;
* BMI (Body Mass Index) ≤ 30 kg/m²;
* With AUFI (type 1 or 2 MRKH syndrome and hysterectomy);
* Informed about the possibility of adoption;
* Compatibility with the donor (ABO group, Human Leukocyte Antigen (HLA) typing);
* Up-to-date vaccinations;
* Able to reach the transplant center in less than 11 hours (applicable only for the "deceased donor" arm);
* Having a parental project that is formulated by a heterosexual couple, by a couple of women or by a single woman;
* Vaginal cup of length greater than or equal to 7 cm.

Inclusion Criteria for a deceased brain-dead uterus donor:

* Any person who is brain dead and who has been duly diagnosed with the following criteria: Female gender;Age ≤ 42 years;Compatibility with the recipient (ABO group, HLA typing).

Inclusion Criteria for a live uterus donor:

* Patient belonging to the family of the recipient (mother, sister, aunt, mother-in-law...) or any person who can prove a stable emotional relationship for more than 2 years with the recipient (paragraphs 1 and 2 of Article L.1231-1 of the Public Health Code);
* Age ≥ 37 years and ≤ 62 years ;
* BMI ≤ 30 kg/m²;
* Having completed all her parenthood plans and no longer having any plans of pregnancy;
* Having had at least one live-born child at term (i.e. after 37 weeks of of amenorrhea);
* Compatibility with the recipient (ABO group, HLA typing);
* Normal suprapubic and/or endovaginal ultrasound or pelvic Magnetic Resonance Imaging (MRI), including uterine (no uterine abnormalities);
* Satisfactory uterine vessels assessed by MRI angio.

Exclusion Criteria for UT recipient:

* Patient with acquired uterine infertility and having had one or more children;
* Non-stable psychological state defined by a clinical psychologist after a qualitative interview;
* Severe co-morbidity;
* Association of severe abnormality with MRKH syndrome other than renal such as a cardiac malformation;
* A single pelvic kidney (urinary malformation that can be associated with MRKH syndrome);
* Pathogenic parental genetic anomaly which may lead to medical termination of pregnancy in the current state of knowledge;
* Diabetes (HbA1c > 6%);
* Disorders of hemostasis: Prothrombin rate <70%;
* Hemoglobin abnormality;
* Existence of hypertension;
* Vaginal reconstruction (neovagina) by digestive segment (colonic plastic surgery or other);
* History of major abdominal or pelvic surgery;
* Known thrombophilia (acquired or constitutional);
* HIV (Human Immunodeficiency Virus), HCV (Hepatitis C Virus), HBV (Hepatitis B Virus), HAV (Hepatitis A Virus), HTLV (Human T-Lymphotropic Virus) serology positive and presence of irreversible communicable infectious diseases;
* Positive vaginal hPV-HR (human Papilloma Virus High Risk) test;
* Signs of chronic renal disease;
* Drug addiction or alcoholism not weaned for more than 2 years or drug addiction or excessive alcohol consumption (> 30 g/day of alcohol) current;
* History of cancer less than 10 years old, cancer under treatment (except in the cancer in situ, or basal cell skin lesion) or diagnosed during the selection process;
* History of pelvic radiotherapy or vaginal brachytherapy regardless of when this irradiation was performed;
* Known psychiatric pathology;
* Active tuberculosis (i.e. under treatment);
* Known or suspected contraindications to one or more of the treatments (active substance or excipient(s)) to be administered for the purposes of the study and/or essential treatment having an interaction/impact with one of the treatments planned by the research;
* Existence of organ dysfunction not compatible with the uterine transplantation protocol;
* History of smoking (defined as consumption greater than 20 packs/year) not weaned for more than 2 years or active smoker.

Exclusion Criteria for a deceased brain-dead uterus donor:

* Initial circulatory arrest of more than 10 minutes;
* Opposition to organ donation (register of refusals) or to uterine removal by a relative of the deceased;
* Chronic and uncontrolled hypertension;
* Absence of uterus (history of hysterectomy or uterine agenesis);
* Presence of uterine pathology;
* Delivery less than 6 months ago or ongoing pregnancy;
* History of several caesarean sections (multi-scarred uterus: more than 2);
* History of major abdominal or pelvic surgery;
* Infection of the sepsis type or uncontrolled infection (bacterial, viral viral, parasitic fungal, active Chagas disease);
* Encephalitis of viral origin or febrile of uncertain origin or meningoencephalitis of unknown origin;
* Risk of Prion disease transmission;
* Presence of an infectious disease: HIV, HCV, HBV, HTLV and presence of irreversible communicable infectious diseases;
* Carrying of human Papilloma Virus High Risk (hPV-HR) class 1 positive in the genital tract if known before transplantation;
* Positive EBV (Epstein-Barr Virus) serology in the donor if the recipient is EBV negative for EBV ;
* Positive pre-transplant virtual crossmatch;
* Donor/recipient ABO final check in the operating room before transplantation positive;
* Drug addiction or alcoholism not weaned for more than 2 years or drug addiction or excessive alcohol consumption (> 30 g/day of alcohol) current;
* History of cancer less than 5 years old, cancer under treatment (except in the cancer in situ, or basal cell skin lesion) ;
* Active tuberculosis (i.e. under treatment);
* History of smoking (defined as consumption greater than 20 packs/year) not weaned for more than 2 years or active smoker.

Exclusion Criteria for a live uterus donor:

* Non-stable psychological state defined by a clinical psychologist clinician after a qualitative interview;
* Severe co-morbidity;
* Diabetes (HbA1c > 6%);
* Hemostasis disorders: Prothrombin rate <70%;
* Hemoglobin abnormality;
* hypertension treated with more than 2 antihypertensive drugs;
* Delivery less than 6 months ago or ongoing pregnancy;
* History of cervical pathology;
* History of recurrent miscarriage syndrome (defined as 3 consecutive consecutive miscarriages);
* History of premature delivery before 36 weeks of amenorrhea;
* History of pre-eclampsia;
* History of caesarean sections;
* History of major uterine surgery;
* History of major abdominal or pelvic surgery;
* Endometrial biopsy and diagnostic hysteroscopy showing an abnormality of the endometrium;
* Known thrombophilia (acquired or constitutional);
* HIV, HCV, HBV, HTLV serology positive and presence of irreversible communicable infectious diseases;
* Positive vaginal hPV-HR (human Papilloma Virus High Risk) test;
* PCR (Polymerase Chain reaction) on HSV (Herpes Simplex Virus) 1/2 positive sample;
* Abnormal vaginal swab;
* Signs of chronic kidney disease;
* Risks of Prion disease transmission;
* Drug addiction or alcoholism not weaned for more than 2 years or drug addiction or excessive alcohol consumption (> 30 g/day of alcohol) current;
* History of cancer less than 10 years old, cancer under treatment (except in the cancer in situ, or basal cell skin lesion) or diagnosed during the selection process;
* History of pelvic radiotherapy or vaginal brachytherapy regardless of when this irradiation was performed;
* Known psychiatric pathology;
* Active tuberculosis (i.e. under treatment);
* Presence of a known thromboembolic risk factor;
* Angio-MRI, CT angiography and/or arteriography revealing an anomaly incompatible with uterine transplantation;
* History of smoking (defined as consumption greater than 20 packs/year) not weaned for more than 2 years or active smoker.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2037-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of uterus transplantation | 6 months after uterus transplantation
  Show a functional uterus validated by the onset of menstruation and maintenance of menstruation 6 months after the uterine transplant has been performed
Security of uterus transplantation | Throughout the UT program
  The number of living children resulting from uterine transplantation relative to the number of recorded complications defined by grade 3 complications of Clavien Dindo (complications of uterine transplant surgery in the post-operative month) and non-reversible complications of immunosuppressants (such as sequelae hypertension, blood disease, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LAVOUE, Principal Investigator — Rennes University Hospital
Locations (1):
- Vincent LAVOUE, Rennes, France